CLINICAL TRIAL: NCT04839991
Title: A Phase 1 Open-Label, Dose Escalation and Expansion Trial to Investigate the Safety, Pharmacokinetics and Pharmacodynamics of CB307, a Trispecific Humabody® T-cell Enhancer, in Patients With PSMA+ Advanced and/or Metastatic Solid Tumours
Brief Title: Study of CB307 in Patients With Advanced and/or Metastatic PSMA-positive Tumours.
Acronym: POTENTIA
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Crescendo Biologics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBT307-1; 2019-004584-46 (EudraCT Number)
Record Dates: First submitted 2021-03-29; First posted 2021-04-09 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Advanced and/or Metastatic Solid Tumours
Keywords: Prostate Specific Membrane Antigen (PSMA); Solid Tumours; Castration-resistant prostate cancer (CRPC); First in Human (FIH); Phase 1 Study; CD137; 4-1BB; Crescendo Biologics; CB307; Humabody®; HSA; Pembrolizumab; KEYTRUDA®

STUDY DESIGN:
Intervention Model Description: Initial dose escalation cohorts followed by dose expansion cohorts consisting of 2 arms, monotherapy and combination therapy cohorts .
Masking Description: Open Label multi center non randomised study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Multi center open label Dose Escalation followed by Cohort Expansion: Part 2A (Experimental): Patients will receive CB307 IV infused every 7 days. Duration of treatment cycle is 21 days. Once the Dose Escalation phase (Part 1) is completed Cohort Expansion phase (Part 2) will begin. Part 2A arm will enrol patients with PSMA+ solid tumours. Treatment will continue until loss of clinical benefit, intolerable toxicity, withdrawal of consent or the study is stopped. Estimated study duration is 20 months.
  Interventions: Drug: CB307
- Multi center open label Dose Escalation followed by Combination Cohort Expansion : Part 2B (Experimental): Patients will receive CB307 IV infused every 7 days in combination with KEYTRUDA® (pembrolizumab) IV infused every 21 days . Duration of treatment cycle is 21 days. Once the Dose Escalation phase (Part 1) is completed Cohort Expansion phase (Part 2) will begin. Part 2B arm will enrol patients with PSMA+ metastatic castration-resistant prostate cancer. Treatment will continue until loss of clinical benefit, intolerable toxicity, withdrawal of consent or the study is stopped. Estimated study duration is 20 months.
  Interventions: Drug: CB307

INTERVENTIONS:
Drug: CB307 — Tri-specific Humabody® targeting CD137, prostate specific membrane antigen and human serum albumin

SUMMARY:
FIH, Phase 1, open-label, multi centre study of CB307, a trispecific Humabody® T-cell enhancer, in patients with advanced and/or metastatic PSMA+ solid tumours to assess safety and tolerability to determine MTD and preliminary RP2D.In addition this study will assess the safety and efficacy of CB307 when given in combination with pembrolizumab (KEYTRUDA®) in patients with metastatic PSMA+ castration-resistant cancer

DETAILED DESCRIPTION:
FIH, Phase 1, open-label, multi centre, non randomised study of CB307, a trispecific Humabody® T-cell enhancer, in patients with advanced and/or metastatic PSMA+ solid tumours (Part 1 & 2A) and patients with metastatic PSMA+ castration-resistant cancer (Part 2B) . The study will consist of a dose escalation phase (Part 1) and a cohort expansion phase (Part 2) which will consist of 2 arms . Part 2 will evaluate safety and preliminary efficacy of CB307 (both as monotherapy and in combination with pembrolizumab) at the MTD or preliminary RP2D as determined in Part 1. Approximately 70 patients will participate in total. Patients will receive either CB307 alone or CB307 with pembrolizumab IV (Part 2B), until loss of clinical benefit, unacceptable toxicity, withdrawal of consent or end of study. The dose escalation may be adapted by the SRC based on clinical experience and safety review.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of understanding the written informed consent
2. Aged at least 18 years
3. Not amenable to standard of care
4. ECOG PS <=2
5. Has documented histologically confirmed diagnosis of PSMA+ advanced or metastatic solid tumours
6. Has radiologically measurable disease per RECIST v1.1 or elevated serum PSA for castration resistant prostate cancer patients with only bone metastasis
7. Adequate organ function

Exclusion Criteria:

1. Subjects with autoimmune disease or regular immunosuppressants
2. Has discontinued from anti-CTLA 4, anti-PD1 or anti-PD(L)1 antibody because of intolerable toxicity
3. Has brain metastasis including leptomeningeal metastasis or primary brain tumour
4. Has current or history of CNS disease
5. Has known active infection
6. Part 2B only - has prior treatment with anti PD(L)1 or anti CTLA4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-06-08 (Actual); Primary Completion 2024-07-25 (Estimated); Study Completion 2024-09-25 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | The nature and frequency of any DLTs during the DLT-monitoring period assessed based on NCI CTCAE v5.0. up to 20 months duration.
  The objective of the study is to assess the safety and tolerability of the study drug CB307 and to determine the MTD (maximum tolerated dose)
Number of participants with treatment-related adverse events with CB307 in combination with pembrolizumab as assessed by CTCAE v5.0 | The nature and frequency of any DLTs during the DLT-monitoring period for participants with combination therapy, assessed based on NCI CTCAE v5.0. up to 20 months duration.
  The objective of the study is to assess the safety and tolerability of the study drug CB307 in combination with pembrolizumab to assess safety and tolerability of the combined treatment regimen

SECONDARY OUTCOMES:
To evaluate clinical efficacy measured as progression-free survival according to RECIST v.1.1 or PCWG3 | Progression-free survival according to RECIST v1.1 or PCWG3 up to 20 months duration; and change from baseline in anti-drug (CB307) antibodies (ADA up to 20 months duration
  To measure how well the treatment succeeds in producing the desired effect.
To evaluate clinical efficacy and duration of response by radiographic progression free survival (rPFS) | radiographic progression free survival up to 20 months duration;
  To measure how well the treatment succeeds in producing the desired effect.
To evaluate anti-tumor response according to RECIST v.1.1 or PCWG3 | anti-tumor response according to RECIST v1.1 or PCWG3 up to 20 months duration;
  To measure how well the treatment succeeds in producing the desired effect.
To measure how the body processes CB307 in the body over time | PK parameters of CB307: data collected at time point 0 at each dosing period up to 20 months duration.
  To evaluate the pharmacokinetic trough levels before administration of CB307
Pharmacokinetic of CB307 T1/2 | Data collected up to 20 months duration.
  To evaluate the pharmacokinetic T1/2 after 3rd dose via IV for multiple dose levels of CB307
Pharmacokinetic of CB307 Tmax | Data collected up to 20 months duration.
  To evaluate the pharmacokinetic Tmax after 3rd dose via IV for multiple dose levels of CB307
To measure Tumour Immune response | Tumor response per RECIST ver 1.1 up to 20 months duration
  To determine the potential of CB307 to produce an immune response and assess the relationship with other outcome measures
Relationship of CB307 to anti tumour response | PSA response defined as a >50% decrease in PSA up to 20 months duration
  To evaluate the preliminary CB307 dose in relationship to activity of changes in tumour

CONTACTS AND LOCATIONS:
Overall Officials: K Hashimoto, Study Director — Crescendo Biologics
Locations (20):
- University of Washington, Seattle, Washington, United States
- Netherlands (5):
  - Antoni van Leeuwenhoek, Amsterdam, North Holland
  - VUMC Research B.V, Amsterdam, North Holland
  - University Medical Center Groningen,, Groningen
  - Erasmus University Medical Center Rotterdam, Rotterdam
  - UMC Utrecht Cancer Center, Utrecht
- Spain (10):
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - hospital clinic de Barcelona, Barcelona
  - hospital de la Sanat Creu i Sant Pau, Barcelona
  - Clinica Universidad de Navarra, Madrid
  - HU Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - NEXT Oncology Hospital Quironsalud Madrid, Madrid
  - HU Virgen de la Arrixaca, Murcia
  - HU Virgen del Rocio - PPDS, Seville
- United Kingdom (4):
  - The Christie NHS Foundation Trust, Manchester, Greater Manchester
  - Royal Marsden Hospital, London, Surrey
  - University College London Hospitals NHS Foundation Trust, London
  - Sarah Cannon Research Institute, UK, London

REFERENCES:
- [Derived] Wilford T, Bartlett PD, Schlag A, Jasaitis L, Pandha H, Pierce AJ, Hughes R. Solving selectivity issues in LBAs: case study using Gyrolab to quantify CB307, a bispecific Humabody in human serum. Bioanalysis. 2024;16(14):757-769. doi: 10.1080/17576180.2024.2365545. Epub 2024 Jul 3. PMID 38957926